CLINICAL TRIAL: NCT02260583
Title: EFFECT OF EXTRACORPOREAL CO2 REMOVAL IN STABLE COPD PATIENTS WITH CHRONIC HYPERCAPNIC RESPIRATORY FAILURE:A PILOT STUDY
Brief Title: Effect of Extracorporeal CO2 Removal in Stable Hypercapnic COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, PRofessor of Respiratory Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 176/2013
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease Patients; Chronic Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- extracorporeal CO2 removal device (Experimental): the patients will be enroll to start a "one shot" session of extracorporeal CO2 removal. The patient will be connected to the device via a double lumen catheter inserted in the femoral vein An ECCO2R device based on a modified continuous venovenous hemofiltration system will be used. Blood flow is driven by a roller nonocclusive pump (0-450 mL/min) through a polypropylene oxygenator ; priming volume, 100 mL; contact surface area, 1.35 m2; maximum blood flow rate, 7 L/min) that is connected to a fresh gas flow source delivering 100% oxygen at a constant rate of 8 L/min. Exiting the oxygenator, blood is driven to a hemofilter.
  Interventions: Device: extracorporeal CO2 device

INTERVENTIONS:
Device: extracorporeal CO2 device — An ECCO2R device based on a modified continuous venovenous hemofiltration system will be used

SUMMARY:
Chronic hypercapnic respiratory failure is common in stable COPD patients in a terminal phase of their disease In an attempt to correct or slow down the rate of rise of PaCO2, long-term noninvasive mechanical ventilation (NIV) has been proposed.

Only very few studies demonstrated the clinical efficacy of NIV. Indeed this technique is not always well tolerated and therefore it may be effective only in a subset of patients The aim of this study is to assess the feasibility and safety of "one shot" extrcorporeal CO2 removal device, in reducing the PaCO2 level

DETAILED DESCRIPTION:
Chronic hypercapnic respiratory failure is common in stable COPD patients in a terminal phase of their disease In an attempt to correct or slow down the rate of rise of PaCO2, long-term noninvasive mechanical ventilation (NIV) has been proposed.

Only very few studies demonstrated the clinical efficacy of NIV. Indeed this technique is not always well tolerated and therefore it may be effective only in a subset of patients Recently extracorporeal CO2 removal have been shown to avoid the need of endotracheal intubation in COPD patients with an episode of Acute Hypercapnic Respiratory Failure In this pilot physiological study we want to assess the safety and efficacy of this technique in reducing the PaCO2 level in those COPD patients with chronic hypercapnic respiratory failure non responding to chronic NIV.

ELIGIBILITY:
Inclusion Criteria:

* COPD ( FEV1/CVF <0.70 post bronchodilation)
* stable PaCO2 >55 mmHg non respondent to long-term NIV (at least one week). This means a decrease in PaCO2 during spontaneous breathing, at least 4 hrs after the termination of NIV, of< 6%
* pH > 7.35
* clinical stability

Exclusion Criteria:

* Mean Arterial Pressure < 60 mmHg
* contra-indication to heparin
* Body Mass Index (BMI) > 30 kg/m2;
* presence of sleep apnea or overall syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
arterial blood gases | 30 days

SECONDARY OUTCOMES:
respiratory rate, dyspnea | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, Principal Investigator — sant'orsola malpighi hospital
Locations (1):
- san'Orsola Malpighi Hospital, Bologna ITALY, Bologna, Italy